CLINICAL TRIAL: NCT05150379
Title: Influence of the Dominance of the Shoulder Stabilized by the Open Latarjet Procedure on the Functional Recovery of the Shoulder at 4.5 Months Postoperatively: Patients Operated on the Dominant Side vs. Patients Operated on the Non-dominant Side vs. Healthy Controls
Brief Title: Influence of the Dominance of the Shoulder Stabilized by the Open Latarjet Procedure on the Functional Recovery of the Shoulder at 4.5 Months Postoperatively.
Acronym: Dom Lat
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: Not yet assigned
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Latarjet; Shoulder Injuries
MeSH Terms: conditions — Shoulder Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dominant side shoulder surgery patients
  Interventions: Other: Different exercises with their shoulders; Behavioral: SI-RSI questionnaire
- Patients operated on the shoulder on the non-dominant side
  Interventions: Other: Different exercises with their shoulders; Behavioral: SI-RSI questionnaire
- Healthy volunteers
  Interventions: Other: Different exercises with their shoulders; Behavioral: SI-RSI questionnaire

INTERVENTIONS:
Other: Different exercises with their shoulders — * Y Balance Test
  * Shoulder rotator muscle isometric maximum strength
  * One handed medicine ball throw
  * Modified Closed Kinetic Chain Upper Extremity Stability Test
Behavioral: SI-RSI questionnaire — French version of Shoulder Instability Return-to-Sport after Injury

SUMMARY:
The aim of this study is to quantify the functional deficits as a function of the dominance of the shoulder stabilized by the open procedure of Latarjet at 4.5 months postoperatively compared to healthy controls.

ELIGIBILITY:
* Patients from two studies : "Reproducibility of functional tests of the shoulder for the return to sport of patients operated on anterior instability of the shoulder "CPP n ° 2018-A03013-52 and "Validation of the S-STARTS composite score to assess the functions of the shoulder and the patient's ability to return to sport after stabilization of the shoulder by the Latarjet procedure (VAL-S-STARTS)" MR3016020520
* healthy volunteers from two studies : "Reproducibility of functional tests of the shoulder for the return to sport of patients operated on anterior instability of the shoulder "CPP n ° 2018-A03013-52" and "Risk factors for shoulder dislocation in rugby players. Predictive validity of the S-STARTS composite score "MR4612110620

Inclusion criteria:

Patients: o patient between 15 and 45 years old

* Occurrence of the injury requiring surgery during a sports activity
* Reduced shoulder instability by the open Latarjet procedure
* Surgery performed by surgeons from the Santy Orthopedic Center (Lyon)
* Inclusion by decision of the surgeon during the visit 4 months postoperatively

Healthy volunteers :

* volunteer between 15 and 45 years old
* Practice a regular sporting activity

Both groups:

* Patient having signed an informed consent
* Subject affiliated or beneficiary of a social security scheme

Exclusion Criteria:

Patient group:

* Contraindication of the surgeon
* Have another pathology in the upper limbs
* Present a constitutional hyperlaxity
* Have stiffness or recurrence of dislocation of the shoulder post-surgery

Healthy volunteers :

* Medical history of upper limb pain / injury within the past 12 months
* Medical history of orthopedic surgery on the upper limbs

Both groups:

* Protected subject: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patient and healthy volunteers between 15 and 45 years old. Patients have an operated shoulder following an injury during a sport activity.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Estimated)
Dates: Start 2021-12-05 (Estimated); Primary Completion 2022-06-05 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
S-STARTS composite score for each participant | 1 hour
  Score between 0 and 21:
  * 0: total functional disability
  * 21: full functional ability

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital privé Jean Mermoz, Lyon, France

REFERENCES:
- [Derived] Rogowski I, Nove-Josserand L, Godeneche A, Colotte P, Franger G, Vigne G, Vieira TD, Blache Y, Neyton L. Functional Deficits After Open Latarjet Procedure and Dominance of the Operated Shoulder: An Analysis of 133 Patients. Am J Sports Med. 2023 Apr;51(5):1277-1285. doi: 10.1177/03635465231156181. Epub 2023 Feb 27. PMID 36847281